CLINICAL TRIAL: NCT03660605
Title: Priming Through Timing. Using Opposing Strategies to Enhance Motor Learning for Improved Gait in Individuals With Parkinson's Disease
Brief Title: Priming Through Timing. Using Opposing Strategies to Enhance Motor Learning for Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-2043
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Parkinson Disease
Keywords: gait; balance; auditory cues
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rhythmic Auditory Stimulation (Experimental): Participants will walk on treadmill to metronome set at 85% of typical cadence, followed by overground walking with metronome set at 115% of typical cadence.
  Interventions: Other: Rhythmic Auditory Stimulation

INTERVENTIONS:
Other: Rhythmic Auditory Stimulation — Participants will complete 6 weeks of walking training (3x/week). During each session, participants will walk on a treadmill for up to 20 minutes (stepping to a metronome at 85% of typical cadence) followed by overground walking for up to 15 minutes (stepping to a metronome at 115% of typical cadence).

SUMMARY:
The purpose of this study is to determine how using auditory cues of a metronome at various frequencies impacts the gait mechanics and balance in people with Parkinson's disease when walking over ground and on a treadmill. We will enroll 10 participants with a diagnosis of Parkinson's disease (Stages 2 or 3). All participants will complete 18 training sessions over 6 weeks and participate in pre- and post-testing of gait and balance.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of Parkinson's Disease (made by movement disorders specialist) will be included in this study. Additional inclusion criteria include: self-reported ability to walk ~6 minutes overground as well as walk on a treadmill for a total of 10 minutes with rest breaks as needed, and be classified as Stage 2, or 3 on the Hoehn and Yahr Scale (Goetz et. al, 2004).

Exclusion Criteria:

* Exclusion criteria include Hoehn and Yahr Stages 1, 4, or 5, uncontrolled cardiorespiratory/metabolic disease (e.g., cardiac arrhythmia, uncontrolled hypertension or diabetes, orthostatic hypertension, chronic emphysema), or other neurological or orthopedic disorders that may affect walking. The investigators will also exclude participants with severe communication impairments, which could impede understanding of the purpose or procedures of the study or an inability to comply with experimental procedures.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
gait speed | one week following conclusion of training
  distance traveled during a 6 minute walk test

SECONDARY OUTCOMES:
cadence | one week following conclusion of training
  number of steps per minute
stride length | one week following conclusion of training
  average length of strides (distance traveled/number of strides)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lewek, PT, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sherron MA, Stevenson SA, Browner NM, Lewek MD. Targeted Rhythmic Auditory Cueing During Treadmill and Overground Gait for Individuals With Parkinson Disease: A Case Series. J Neurol Phys Ther. 2020 Oct;44(4):268-274. doi: 10.1097/NPT.0000000000000315. PMID 32459723